CLINICAL TRIAL: NCT06000462
Title: The Effect of Sodium Glucose Co-transporter 2 Inhibitor (dapagliflozin) on Weight Loss in Non-diabetic Adults with Obesity: Triple-blinded, Randomized, Placebo-controlled Trial.
Brief Title: The Effect of Dapagliflozin on Weight Loss in Obese Adults Without Diabetes
Acronym: DAPA-ANDO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oman Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Thuraiya Malik Al Harthi, Epidemiologist, Oman Ministry of Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OmanMOH
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Dapagliflozin Adverse Reaction; Weight Loss; Effect of Drug
Keywords: Sodium glucose co transporter inhibitor 2; Dapagliflozin; weight reduction; obesity; young adult; SGLT2I; weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — dapagliflozin; Metformin; Disulfiram

STUDY DESIGN:
Intervention Model Description: Triple-blind, parallel groups, randomized, placebo control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To blind the care providers, investigators, and participants,150 packs of medication labelled from 1 to 150 numbered randomly from 1-150 (but this depends on number of patients who did not respond to run in period intervention), 50 each containing either 10 mg dapagliflozin or 1000mg metformin or the placebo. The label on the pack only has the serial number but the pharmacist (who is not part of this study) has the code of what each bottle contains and that is kept safely and confidentially (Hard copy and multiple soft copies in safe custody). Participants are numbered serially according to recruitment, and each gets the correspondingly numbered bottle (which has been previously randomly assigned by the pharmacist).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dapagliflozin (Experimental): 10 mg strength will be used in this study. The drug is usually taken orally once a day, preferably in the morning. The participants will be using the medication for 32 weeks only, then continue follow up for another 16 weeks (off drug therapy) with behavior weight management program only. The patients will be informed from the beginning of the study with the general side effects of medication (patient information sheet) that should be reported if experienced.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Metformin (Active Comparator): 1000 mg strength will be used once daily dose taken orally. Medication will be provided randomly to the patient according to the corresponding number. The patients are informed to declare any experienced side effects that has been stated in the patient information sheet without informing the name of drugs.
  Interventions: Drug: Metformin 1000 mg (ttd)
- Placebo (Placebo Comparator): receive a non-medicated pill that has no therapeutic effect, once daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Mentioned in detailed description.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Metformin 1000 mg (ttd) — A dose of 1000 mg, PO, once daily, given over 8 months period
  Other Names: Glucophage
  Arms: Metformin
Other: Placebo — a non-medicated pill will be used as a placebol
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of a drug named dapagliflozin (tested drug) on weight loss in young adults aged between 18 and 40 years with obesity who are not diagnosed with diabetes.

The main questions this study aims to answer are:

* How much weight in average can people loose with the use of tested drug compared to 2 other comparator drugs: metformin and placebo (non-medicated pill)?
* What is the effect of using tested drug on other parameters used to assess metabolic disease including blood pressure, cholesterol and sugar levels, and mental health?
* How frequent are the side effects from using the tested drug compared to the comparator drugs? Participants will go through a 6-month program of physical activity and diet and measure their weight progress (Run in period). Those who do not achieve the target weight reduction will be randomly assigned to any of the three drug groups, either testes drug group, comparator 1 (metformin), or comparator 2 (placebo).

DETAILED DESCRIPTION:
Background Obesity is a disease, generally defined as a body mass index (BMI) ≥ 30 kg/m2,1 is a global issue that continues to grow at an alarming rate, imposing serious threat to individuals, public health, and the economy. The prevalence of overweight and obesity has tripled since 1975, with 1.6 billion overweight adults and 650 million obese adults, according to World Health Organization report.2 In Oman, non-communicable diseases (NCDs) represent a major burden on healthcare system at which 185.75 deaths per 100,000 population are attributed to NCDs.3 Obesity is an independent risk factor for most NCDs, adding to disease morbidity and mortality. According to a national survey conducted in 2017, the prevalence of obesity and overweight were 30.7% and 66.1%, respectively, with higher prevalence in females compared to males.4 The Look AHEAD trial revealed that losing 5% to 10% of body weight through diet and exercise alone has been associated with reduced risk of cardiovascular disease in obese and overweight adult patients.5 Whilst healthy lifestyle is the mainstay for obesity management, there is a growing interest over pharmaceuticals that support weight loss and prevent metabolic complications.

The US Food and Drug Administration (FDA) approved five drug therapies to treat obesity, namely orlistat, phentermine/topiramate, lorcaserin, naltrexone/bupropion, liraglutide, and recently saxenda,6 while the European Medicines Agency (EMA) supported three drug therapies, orlistat, bupropion/naltrexone and liraglutide.7 Several anti-diabetic drugs have been authorized for weight loss even for patients without diabetes.8 Sodium glucose cotransporter 2 inhibitors (SGLT2i) including empagliflozin, dapagliflozin and canagliflozin are classes of hypoglycemic agents that have been studied in both human and animal models to measure their glycemic and metabolic effect. These drugs reduce plasma glucose levels by inhibiting the sodium glucose cotransporter 2, located in the proximal tubule of the kidney, leading to increased urinary glucose excretion and a reduction in plasma glucose levels in patients with type 2 diabetes mellitus (T2DM).8-11 This mechanism of action was found to lower the risk of hypoglycemia, with additional benefits of weight loss, reductions in blood pressure, cardiovascular (CVD), and chronic kidney disease risk (CKD). 8, 12, 13 The drugs are prominent in most recent guidelines for the management on T2DM and are particularly recommended when, in addition to glucose lowering, there is a compelling need to reduce body weight.14 Weight reduction via behavior change and maintaining healthy lifestyle is the first line and cost-effective treatment for obesity. According to the US Preventive Services Task Force, all adults aged 18 years or above should be screened for obesity and intensive behavior intervention to be given for weight loss,15 with at least one session per month for at least three months.16 Body mass index (BMI) is a key indicator for weight assessment; however waist circumference may be an acceptable alternative in people with central obesity because BMI may not account for the cardiovascular risk of central adiposity.17

Dapagliflozin is a highly selective SGLT2i that blocks the reabsorption of 80% - 90% of the glucose filtered by the glomerulus. It is an oral medication with three different dose strengths; 2.5 mg, 5mg, 10 mg once daily, in addition to the combination formula with metformin; dapagliflozin/ metformin, with strength of 2.5mg/1000mg, 5mg/500mg, 5mg/1000mg, 10mg/500mg, and 10mg/1000mg. Several RCTs have shown its effectiveness on glycaemic control, weight loss, and blood pressure in patients with T2DM, in addition to the cardiovascular and renal protection.24 A randomized placebo control trial (RCT) that enrolled 534 patients with T2DM on preceding metformin treatment investigated the effectiveness of dapagliflozin 2·5 mg, 5 mg, and 10 mg per day dose versus placebo, over 24 weeks. There was a dose dependent reduction in HbA1c in patients treated with dapagliflozin, with a reduction of 0·84% in patients assigned to a maximum dose of 10 mg per day compared with a reduction of 0·3% in the placebo group, at the end of study period. Mean HbA1c had decreased by -0·30% (95% CI -0·44 to -0·16) in the placebo group, compared with -0·67% (-0·81 to -0·53, p=0·0002) in the dapagliflozin 2·5 mg group, -0·70% (-0·85 to -0·56, p<0·0001) in the dapagliflozin 5 mg group, and -0·84% (-0·98 to -0·70, p<0·0001) in the dapagliflozin 10 mg group.25 The trial also showed no apparent changes in fasting lipid profiles, apart from greater mean increases in HDL cholesterol (1·8-4·4% vs 0·4%) and decreases in triglycerides (-2·4% to -6·2% vs 2·1%) compared with placebo.25 Treatment with dapagliflozin was not superior to placebo in reducing the risk of major adverse cardiovascular events but lowered the risk of hospitalization due to heart failure or death from CVD (hazard ratio: 0.83; 95% CI, 0.73 to 0.95; P=0.005).26 In patients with established chronic renal disease with an estimated glomerular filtration rate (eGFR) of 25 to 75 ml per minute per 1.73 m2 of body-surface area and/ or urinary albumin-to-creatinine ratio of 200 to 5000) who received dapagliflozin 10 mg a day, showed a significantly lower risk for sustained decline in the estimated eGFR of at least 50%, end-stage kidney disease, or death from renal or cardiovascular causes than with placebo. The hazard ratio for renal dysfunction or death from renal causes was 0.56 (95% CI, 0.45 to 0.68; P<0.001) in dapagliflozin compared with placebo and a hazard ratio 0.71 (95% CI, 0.55 to 0.92; P=0.009) for death from cardiovascular causes or hospitalization for heart failure.27 In patients with mild to moderate chronic kidney disease of diabetes, no alterations in mean renal function measures, including serum creatinine concentration, were reported.28 The most common side effects of dapagliflozin were urinary and genital infection, 29 besides headache, backpain, and diarrhea.30 An analysis of published data from 12 RCTs, included 3152 patients who received dapagliflozin 2.5 mg, 5 mg, or 10 mg as monotherapy or add-on treatment, and 1393 placebo-treated patients, showed that the diagnosis of infection were reported in 3.6%, 5.7%, 4.3%, and 3.7%, respectively. However, most infections were treated and responded to antimicrobial therapy. Discontinuations due to urinary tract infection were rare: 8 (0.3%) dapagliflozin-treated patients and 1 (0.1%) placebo-treated patient.30 Most studies were in patients with diabetes who are at risk of asymptomatic bacteriuria and pyelonephritis in combination with dysfunction of the urinary tract compared with people without diabetes, the fact that further studies with longer observation period are required to confirm that infection is related to the drug and not diabetes status.31 In fact, it has been found that the frequency of serious adverse effects including urinary and genital fungal infection from dapagliflozin were comparable to placebo in patients with T2DM.30 Dapagliflozin and obesity management Obesity and T2DM are intrinsically linked with multiple shared pathology, besides being associated with increased risk of multiple comorbidities.32 The weight loss observed with SGLT2i is thought to be due to fluid loss, reduction in lean body mass, and thereafter loss of calories via increased urinary glucose excretion. Dapagliflozin was found to improve adipocyte function by lowering inflammatory markers, C-reactive protein and increasing adiponectin besides lowering glycated hemoglobin and body weight, however evidence was inconclusive due to small sample size.33 Animal based trials are still ongoing to provide evidence of actual mechanism of weight loss with SGLT2i. Modest body of evidence have shown the effectiveness of dapagliflozin in causing clinically significant reductions in body weight.34 A double-blind placebo-controlled study of 182 patients with T2DM treated with dapagliflozin 10mg a day versus placebo (added on metformin) over 102 weeks showed reductions in HbA1c by -0.3%, weight by -4.54 kg, waist circumference by -5.0 cm and fat mass by -2.80 kg without increases in rate of hypoglycemia, in former drug compared with later placebo. In addition to that, no significant changes from baseline in bone density or markers of bone turnover, compared with placebo. The frequency of patients with at least one adverse event (mainly urinary and genital infections) were comparable; 71.4% in the dapagliflozin and 69.2% in placebo group by week 102. 35 Another RCT compared the metabolic effect of dapagliflozin versus placebo on high density lipoprotein (HDL-C) over 16 weeks of treatment, showed reduced HbA1c by 0.9% and body weight by 3.1 kg, mainly attributable to reduction of body water and lean mass, without evidence of improving HDL-cholesterol.36 Treatment with dapagliflozin 5 mg/day over 24 weeks showed a decrease in total body weight of 2.9kg (3.9%). Furthermore, there was a decrease in serum alanine aminotransferase and γ-glutamyl transpeptidase levels and a significant decrease in controlled attenuation parameter (CAP)- a measure of liver stiffness and fibrosis from 314 ± 61 to 290 ± 73 decibel dibutyryl (dB)/m (P = 0.0424), concluding that dapagliflozin might improve liver steatosis in patients with type 2 diabetes and NAFLD. However, the possibility that a reduction in body weight or visceral adipose tissue by dapagliflozin may be associated with a decrease of liver steatosis or fibrosis, cannot be excluded.37 A small, prospective study of 26 patients with T2DM who received dapagliflozin 5mg/day over 12 weeks showed a 23.8% loss of lean body mass but modest weight loss of 2.5 Kg.36 A randomized double blind placebo control trial showed that empagliflozin monotherapy at doses of 10 mg and 25 mg for ≥76 weeks was well tolerated and led to sustained reductions in glycated hemoglobin (HbA1c) and weight compared with placebo.37 The glucose-dependent mechanisms of action of SGLT2-i comes with low risk of hypoglycemia, particularly when not used with sulphonylureas or insulin.38 Several studies have been undertaken to evaluate and measure the effectiveness of SGLT-2i in managing obesity in diabetic and non-diabetic patients, however evidence is inconclusive and necessitates further high-quality trials to assess the long-term outcomes of this drug that is administered orally, once daily dose, with expected low risk of severe adverse events.

The trial will evaluate the efficacy and safety of dapagliflozin compared to metformin and placebo in weight loss management in young adults with obesity, who are not yet diagnosed with diabetes.

Methods:

Study design:

All subjects will be prescribed a structured monitored and tailored program from the beginning of the 24-week run-in period before randomization to drug therapy.

Patients who do not respond to the structured lifestyle program (not losing 5-10% of weight) will be randomized to any of the three arms: placebo, metformin, or dapagliflozin.

After randomization, participants will go through 48-week double-blind, randomized, parallel-group, placebo-controlled, trial. In the first 32 weeks, subjects will be randomized 1:1:1 to receive either dapagliflozin 10 mg or metformin 1000 mg or placebo. The randomization will be stratified according to age and metabolic parameters. After 32 weeks drugs will be discontinued and patients will be followed for another 16 weeks after end of drug therapy "off-study-drug follow-up period" to assess effect maintenance and any evidence of rebound, as well as to monitor post-treatment safety.

Trial interventions:

- Run- in period:

1. Behavioral weight management program alone:

   Physical activity:

   At baseline visit, the participants will be given a physical activity prescription written by the family physician/ endocrinologist in obesity clinic to guide type and frequency of exercises. Participants will be enrolled in a structured program for physical activity in a fitness gym that is well-known of high fitness, health, and safety standards throughout the study period - 24 (run-in) and 48 (post randomization) weeks. A list of participant names will be given to a prespecified branch according to patients' location preference. Each gym should nominate fitness instructors to monitor the way workouts are done by the participants. A logbook approach will be used to ensure adherence by patients and instructors, in which patients must submit to the care provider every time they visit the clinic on their appointment. The logbook will include information regarding date, time, type of exercise, duration of exercises, progress. In case any participant missed more than one class, the instructor is expected to call for a reminder and reschedule for the missing session. Type of exercises will include muscle strengthening and aerobic exercises using machines. The participant is expected to complete 75 to 150 minutes for muscle strengthening and 150 - 300 minutes for cardio-based exercises per week, to achieve the World Health Organization recommendation for physical activity, hence, at least 4 sessions of 30 minutes in each per week, might be a target.

   Nutrition counselling clinical nutritionist will be involved in providing proper dietary and behavior modification counselling to all study participants and maintain schedule follow ups later. Patients will be seen at baseline, 24 weeks, 48 weeks from baseline. The nutritionists have been trained on motivational interview skills as part of their professional development, hence motivation and encouragement care will be provided during the dietary counselling sessions. The dietary plans will mainly focus on calorie reduction rather than specific dietary composition of macronutrients to make it simple, without overwhelming patients and ensure good adherence. A deficit of at least 500 kcal per day can be achieved with intake of 1,200 to 1,500 kcal for women and 1,500 to 1,800 kcal for men. Although different diets with similar caloric intake can result in comparable weight loss, a higher-quality diet of nutrient-dense foods (e.g., vegetables, fruits, whole grains) that are rich in fiber, vitamins, and minerals will produce greater results. Dieticians will follow the general guidance from Dietary Guidelines for Americans 2015 - 2020 that reinforces the need for healthier food and beverage choices by consuming nutrient-dense foods from all food groups and limiting intake of added sugars, saturated fats, and sodium. In addition, intermittent fasting schedule will be incorporated into the dietary regime.

   Behavior modification counselling Motivational interview will be the main technique used to encourage behavior change and adherence to healthy lifestyle including physical activity and low-calorie diet. The technique includes 1. Asking permission to discuss behavior change, 2. Showing empathy throughout discussion, 3. Using scale of motivation and confidence, 4. Enquiring about the chosen scores, 5. Exploring barriers to change, 6. Exploring pros and cons of behavior change. 7. Listening to change talk "where the patient takes the ownership to generate ideas and ways" and reinforce it. The psychologists will provide comprehensive counselling at baseline and 12 weeks from baseline, besides the scheduled counselling that will be given by dieticians throughout the scheduled follow ups.
2. Pharmacotherapy

Recruitment of patients:

Recruitment will take place over a 6-month period in the primary care health centers by the trial investigators. Patients fulfilling the inclusion criteria will be provided with a participant information sheet about the study by the project officers and patients showing interest will be given a consent sheet to confirm participation and adherence to study conditions in written. Participants will be involved in 24 weeks (6 months) run in period to provide them with a comparable behavior modification and healthy lifestyle program in their health centers before randomization to ensure homogeneity and patient safety as drug of interest is used off-label. Appointments will be given to all participants to attend the obesity clinic for baseline measures and to receive care in polyclinics. Recruitment will be monitored on a monthly basis and efforts to reduce loss to follow-up will be made. Participants not attending their appointment will be called to consider rescheduling their appointments.

Key randomization criteria:

* BMI corresponding to 30-35 kg/m2 for adults by international cut-off points (for diagnosis of obesity).
* Compliance with run-in procedures and visit schedule (during the period between screening and randomization) as judged by the investigator.

Randomization and allocation concealment After recruitment of eligible participants, computerized number generator will be used to generate random identification of study arms and patients, stratified according to age, gender, and metabolic parameters. The allocation would be 1:1:1to each arm of the study group. An independent healthcare professional "most probably a nurse" who is not part of the study team will lead the allocation concealment of the randomized groups who will also be concealed from the study arms. The arms will be coded A, B, C and only independent nurses will be aware of these codes that are saved and registered electronically.

Ensure patient safety:

Any study participant is noticed to have side effects that warrants the clinician to know with certainty, the medication he/she has been receiving will be identified through the pharmacists who have the key to the codes and will be asked to reveal the medication given to that patient. The treating physician will manage the patient with this knowledge. If several patients show side effects and the code shows them to be in the same treatment arm, a decision can then be made to discontinue that arm or stop the study (as per the severity or risk of continuing the study) all these safety features can be built into the study.

Sample size:

To demonstrate a between groups difference of 5kg in body weight over 3 months from baseline, that would be detected at a power of 80%, with significance level of 5%, and a standardized difference of 0.700 gm (i.e., 0.394 of a standard deviation can be detected), the minimum required sample size is 300 (75 in each arm). With an attrition rate of 20% and a recruitment rate of 70% the required sample size is 500 (125 in each arm). However, due to patient safety issue related to using a drug off-label, a sample size of 150 will be used in this study.

Data monitoring/ management Every two weeks, a research nurse will collect and process electronic enrollment and randomization data, which will then be stored, reviewed, and shared as anonymous files. Follow-up data will be obtained and updated quarterly, while real-time monitoring will be conducted for deaths. Every six months, a batched process will be used to assess and make decisions on adverse events in patients who have exceeded the 6-month observation period. An independent statistician, who is not privy to the study's unblinded data, will analyze and compile reports for the Drug safety team pharmacist every six months. The study investigators will conduct annual audits of site data collection and procedures, ensuring that no outcome or endpoint information is shared with clinical sites. Enrolment and follow-up statistics will be accessible in a secure, password-protected section of the trial's website.

Statistical analysis The intra group and intergroup differences in percentage of usual weight change and mean weight and BMI will be calculated. It will generally be presented by two-sided confidence intervals (CIs) with a confidence level of 95%. Superiority will be claimed if the two-sided p-value is less than 5% and the treatment estimate favors dapagliflozin arms. If the upper limit is below 0, superiority of dapagliflozin against metformin and placebo can be concluded.

• Analysis of outcomes The full analysis set (FAS) will be used in the analysis of the efficacy endpoints. For the safety endpoints, the safety analysis set (SAS) will be used.

FAS: includes all randomized subjects who have received at least one dose of trial product and have any post-randomization data. The statistical evaluation of the FAS will follow the intention-to-treat (ITT) principle and subjects will contribute to the evaluation "as randomized".

SAS: includes all subjects exposed to at least one dose of trial product. Subjects in the SAS will contribute to the evaluation "as treated".

Before data are locked for statistical analysis, a blinded review of all data will take place. Any decision to exclude a subject or single observation from the statistical analysis is the joint responsibility of principal investigator and co investigators. Exclusion of data from analyses will be used restrictively and normally no data should be excluded from the FAS. The subjects or observations to be excluded, and the reasons for their exclusion must be documented and signed by those responsible before database lock. The subjects and observations excluded from analysis sets, and the reason for this, will be described in the clinical trial report Handling of missing values Missing data in the main analysis will be handled by the following multiple imputation (MI) method. A pattern mixture model approach is applied where withdrawn subjects or treatment discontinued subjects without a follow-up visit are assumed to respond as if treated with placebo for the entire trial. Multiple copies (100 copies) of the full dataset will be generated by imputing missing values based on estimated parameters for the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-40 mg/kg2 for adults by international cut-off points (for diagnosis of obesity)
* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Stable body weight during the previous 90 days before screening (<5 kg self-reported weight change)
* History of failing to lose sufficient weight with lifestyle modification as judged by the investigator and documented in subject's medical record.

Exclusion Criteria:

* Type 1 or type 2 diabetes mellitus (T1DM)
* Subjects with secondary causes of obesity (i.e., hypothalamic, genetic, or endocrine causes)
* Treatment with medications within 90 days before screening that, that are used in obesity treatment including pramlintide, orlistat, zonisamide, topiramate, lorcaserin, phentermine, bupropion, naltrexone, glucagon-like peptide-1 (GLP-1) receptor agonists, or metformin (used as treatment for obesity)
* On anti-diabetic treatment
* Patients with impaired kidney function including persistent eGFR <= 45 and albuminuria
* Patients with peripheral vascular disease
* Patients with recurrent urinary tract infection or fungal infections within 12 months before screening
* History of major depressive disorder within 2 years before screening
* History of cardiopulmonary diseases that prevents from physical activity
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in inter-arms percent of subjects achieving ≥5% reduction in baseline weight | 32 weeks post randomization
  we will measure the percentage change of weight in terms of achieving 5 or more and compare it with other arms
Inter-arms differences in mean BMI, waist circumference, waist hip ratio, body weight (kilogram, kg), Body fat (%), and Muscle mass (%) | 32 weeks post randomization
  we will measure the intra-group mean difference from baseline and then compares the intergroup mean difference.

SECONDARY OUTCOMES:
Inter-arms group mean difference in metabolic parameters, depression, anxiety | 32 weeks post randomization
  we will measure the intra-group mean difference from baseline and then compare the intergroup mean difference.
Frequency of adverse event from dapagliflozin | 32 weeks post randomization
  We will monitor patients for the development of any signs or symptoms suggestive of side effect and calculate the prevalence. The prevalence rate will be compared between the study arms

CONTACTS AND LOCATIONS:
Overall Officials: Thuraiya Al Harthi, Masters, Study Director — Oman MoH
Locations (1):
- Bawsher Health Center, Bawhser, Muḩāfaz̧at Masqaţ, Oman

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participants data with regards to amount of weight loss and changes in metabolic parameters after receiving the intervention
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 24 months
Access Criteria: principal investigator Research assistant Care providers Statistician

REFERENCES:
- [Background] Lin X, Li H. Obesity: Epidemiology, Pathophysiology, and Therapeutics. Front Endocrinol (Lausanne). 2021 Sep 6;12:706978. doi: 10.3389/fendo.2021.706978. eCollection 2021. PMID 34552557
- [Background] WHO. Obesity and Overweight. 2018. 23 Feb 2020. Contract No.: https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight.
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Al-Mawali A, Jayapal SK, Morsi M, Al-Shekaili W, Pinto AD, Al-Kharusi H, Al-Harrasi A, Al-Balushi Z, Idikula J. Prevalence of risk factors of non-communicable diseases in the Sultanate of Oman: STEPS survey 2017. PLoS One. 2021 Oct 28;16(10):e0259239. doi: 10.1371/journal.pone.0259239. eCollection 2021. PMID 34710161
- [Background] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- [Background] Food U, Administration D. FDA Approves New Drug Treatment for Chronic Weight Management: First Since 2014. Washington, DC Center for Drug Evaluation and Research. 2021.
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Background] DeFronzo RA, Davidson JA, Del Prato S. The role of the kidneys in glucose homeostasis: a new path towards normalizing glycaemia. Diabetes Obes Metab. 2012 Jan;14(1):5-14. doi: 10.1111/j.1463-1326.2011.01511.x. PMID 21955459
- [Background] Liu XY, Zhang N, Chen R, Zhao JG, Yu P. Efficacy and safety of sodium-glucose cotransporter 2 inhibitors in type 2 diabetes: a meta-analysis of randomized controlled trials for 1 to 2years. J Diabetes Complications. 2015 Nov-Dec;29(8):1295-303. doi: 10.1016/j.jdiacomp.2015.07.011. Epub 2015 Jul 21. PMID 26365905
- [Background] Gallo LA, Wright EM, Vallon V. Probing SGLT2 as a therapeutic target for diabetes: basic physiology and consequences. Diab Vasc Dis Res. 2015 Mar;12(2):78-89. doi: 10.1177/1479164114561992. Epub 2015 Jan 23. PMID 25616707
- [Background] Michel MC, Mayoux E, Vallon V. A comprehensive review of the pharmacodynamics of the SGLT2 inhibitor empagliflozin in animals and humans. Naunyn Schmiedebergs Arch Pharmacol. 2015 Aug;388(8):801-16. doi: 10.1007/s00210-015-1134-1. Epub 2015 Jun 26. PMID 26108304
- [Background] Baker WL, Smyth LR, Riche DM, Bourret EM, Chamberlin KW, White WB. Effects of sodium-glucose co-transporter 2 inhibitors on blood pressure: a systematic review and meta-analysis. J Am Soc Hypertens. 2014 Apr;8(4):262-75.e9. doi: 10.1016/j.jash.2014.01.007. Epub 2014 Jan 26. PMID 24602971